CLINICAL TRIAL: NCT02161081
Title: Adenosine-induced Stress Myocardial Perfusion Imaging With Dual-source 128-slice CT: a Study on the Comparison of Diagnostic Performance of Dynamic Scanning Protocols
Brief Title: A Study on Improved Dynamic Myocardial Perfusion With Less Effective Radiation Dose in CT (SIMPLE CT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SMC2011-05-032-023
Record Dates: First submitted 2014-03-31; First posted 2014-06-11 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2014-03

CONDITIONS: Myocardial Ischemia
Keywords: Myocardial ischemia; Coronary artery disease; Myocardial CT perfusion; Modified scan protocol; Diagnostic performance; Radiation dose
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myocardial CT perfusion (21-second) (Experimental): A total of 60 symptomatic patients will be randomized to dynamic CT perfusion protocol with 21-second scan duration.
  Interventions: Procedure: Myocardial CT perfusion
- Myocardial CT perfusion (30-second) (Active Comparator): A total of 60 symptomatic patients will be randomized to dynamic CT perfusion protocol with 30-second scan duration.
  Interventions: Procedure: Myocardial CT perfusion

INTERVENTIONS:
Procedure: Myocardial CT perfusion — Adenosine-stress dynamic myocardial CT perfusion using 128-slice dual-source CT

SUMMARY:
Among the current myocardial CT perfusion techniques, dynamic CT perfusion technique is most advantageous in obtaining information on myocardial blood flow and volume. However, dynamic CT perfusion technique involves higher radiation dose than static CT techniques. Patients have to take a breath hold during 30 seconds with current dynamic CT perfusion protocol. If patients cannot hold their breath, anterior or inferior myocardium might be excluded due to limited scan coverage of a 128-slice dual-source CT scanner.

Reduction of scanning duration of dynamic CT perfusion may not only reduce radiation exposure, but also make patients more comfortable. Therefore, the investigators intended to propose a modified scan protocol with shorter scan duration and compare diagnostic accuracy of a modified scan protocol with the current scan protocol.

DETAILED DESCRIPTION:
The aim of this study is to compare the diagnostic performance of adenosine-stress dynamic myocardial CT perfusion using a reduced dynamic scan duration with perfusion protocol of 30-second scan duration for the detection of myocardial perfusion defect and significant coronary artery stenosis.

This trial is a single center, prospective, randomized trial designed to compare diagnostic performances and radiation doses between two protocols with 30-second or 21-second dynamic scan durations. A total of 120 symptomatic patients will be randomized to dynamic CT perfusion protocols with 30-second or 21-second scan duration. They will also undergo 1.5-T MRI and invasive coronary angiography as reference standards for the assessment of myocardial perfusion and coronary artery stenosis. The primary end point of the study is to compare diagnostic performances between two CT protocols of dynamic CT perfusion. The secondary endpoint of this study is to compare radiation doses and image qualities of two scan protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women patients, with age ranging 30-80.
2. Known or suspected coronary artery disease who are supposed to undergo invasive coronary angiography
3. Patients who are willing to sign the informed consent form

Exclusion Criteria:

1. Contraindication of CT

   * Known allergy to iodinated contrast media or history of contrast-induced nephropathy
   * Decreased renal function: elevated serum creatinine (>1.5 mg/dl)
   * Severe arrhythmia: atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third degree heart block)
   * Severe thyroid disease
   * Homocystinuria
   * History of asthma
   * Hypersensitivity to adenosine
   * Severe obstructive lung disease
   * Intake of caffeine or xanthine-containing compounds within the last 48 hours
2. Contraindication of MRI

   * Claustrophobia
   * Metallic hazards
   * Pacemaker implant
   * eGFR (estimated glomerular filtration rate) <30 ml/min
   * Clipping for aneurysm (stainless steel clips), neurostimulator, cochlear implant.
3. Unstable or uncooperative patients
4. Limited life expectancy due to cancer or end-stage renal or liver disease
5. Evidence of severe symptomatic heart failure (NYHA Class III or IV)
6. Acute myocardial infarction, hypertrophic cardiomyopathy, dilated cardiomyopathy, coronary artery bypass surgery, or other cardiac surgery
7. Women with positive pregnancy tests

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) of CT perfusion for detection of perfusion defects : 30-second scanning protocol versus 21-second scanning protocol | When all randomized patients underwent CT scanning (A total of 120 symptomatic patients will be randomized to dynamic CT perfusion protocols with 30-second or 21-second scan duration.)
  There were no significant differences in the diagnostic performances between two CTP protocols with different scan duration.

SECONDARY OUTCOMES:
Effective radiation dose for each component of the CT examination is calculated as the product of the dose-length product multiplied by a conversion coefficient of 0.014 (mSv/[mGycm]). | up to 1 week after each patient underwent CT scanning
  CTP with shorter scan duration resulted in a 23% reduction of radiation dose compared with 30-second scan protocol

CONTACTS AND LOCATIONS:
Overall Officials: Yeon Hyeon Choe, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea